CLINICAL TRIAL: NCT01293864
Title: Structural Analysis of Human Tissue
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trials study
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00002154
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2015-12

CONDITIONS: Cutis Laxa
Keywords: structural analysis, diffusible proteins, glycosaminoglycans
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Abdominal tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The object of this study is to analyze fresh human skin samples using several up-to-date technologies to get parameters on the mechanical, biochemical and structural distribution of the main components of the capillary-tissue unit.

Our working hypothesis is that both structural components of the dermis are not evenly distributed along parallel planes. The investigators further hypothesize the the distribution patterns determine functional and mechanical differences along dermal layers.

DETAILED DESCRIPTION:
Background The skin is a large organ that participates in many protective and homeostatic processes. The functions of the skin can be roughly divided into systemic and local ; both are interrelated but relationships are poorly understood and studying them requires a multiscale approach. Particularly, for the local responses that are mediated by activation of proteolytic and signaling pathways such as coagulation and inflammation, the relevant scale corresponds to the micrometer and nanometer dimensions of cells and macromolecules, respectively. There is very little information on the physicochemical characteristics of the skin at these scales.

Objective The investigators propose to analyze fresh human skin samples using several up-to-date technologies to obtain parameters on the mechanical, biochemical and structural distribution of the main components of the capillary-tissue unit.

Hypothesis/Rationale Our working hypothesis is that both structural components of the dermis, such as glycosaminoglycans, and key mediators of homeostatic pathways, such as the procoagulant tissue factor are not evenly distributed along parallel planes. The investigators further hypothesize that the distribution patterns determine functional and mechanical differences along dermal layers.

Methods Using a dermatome, human skin will be dissected along planes parallel to the epidermis into several layers each approximately .0012mm thick. The layers will be analyzed with respect to composition of diffusible proteins and glycosaminoglycans; subjected to high resolution MRI and AFM scanning; and evaluated for swelling rate and equilibrium swelling pressure.

Significance This study will provide new information on material characteristics and functional structure of the human skin at resolutions relevant to the macromolecular and cellular processes that mediate local responses to injury and maintain local homeostatic mechanisms. The data will be further processed to obtain realistic parameters that are needed to develop predictive models of the skin capillary tissue unit. These models will bring new and deeper understanding on skin physiology and pathology and will aid in the discovery and testing of new preventive and therapeutic approaches targeting dysfunctions of the local homeostatic balance in the skin. Potentially, by exploiting the versatility of mathematical simulations in the skin model, the findings will also be applicable to other tissue organs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, male or female , between the ages of 18 to 65 years of age, who will be having surgery to remove excess skin from the abdominal area by surgeons in the Department of Plastic & Reconstructive Surgery

Exclusion Criteria:

* Subjects younger then 18 years of age or older than 65 years of age, and are not having excxess skin surgically removed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of patients who are being seen in the Plastic & Reconstructive Surgery Clinic for surgical removal of excess abdominal skin (abdominoplasty).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morykwas, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Department of Plastic & Reconstructive Surgery, Winston-Salem, North Carolina, United States